CLINICAL TRIAL: NCT04988789
Title: Evaluation of Paclitaxel Coated Balloon in the Treatment of Dialysis Access Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/2320
Record Dates: First submitted 2021-07-25; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Dialysis Access Malfunction; Kidney Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Paclitaxel Drug Coated Balloon — Failing AVF/AVGs treated with Paclitaxel Drug Coated balloons are captured in this database

SUMMARY:
Recent studies of paclitaxel DCB in the treatment of stenosis at dialysis vascular access have shown promising results. Paclitaxel, an anti-proliferation drug, is released during balloon inflation and potentially improve primary patency by slowing down NIH effect. However, meta-analysis have suggested that the use of paclitaxel in lower limbs have increased risk of death in patients. The effect of paclitaxel DCB on dialysis access however remains unknown. Hence, we aim to set up a database to track long-term treatment outcomes of patients treated with Paclitaxel DCB at SGH for their stenosed dialysis access

ELIGIBILITY:
Inclusion Criteria:

* All patients above 21 that is undergoing AVF/AVG fistuloplasty with paclitaxel DCB at SGH is included

Exclusion Criteria:

* All patients below 21

Ages: 21 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients above 21 that is undergoing AVF/AVG fistuloplasty with paclitaxel DCB at SGH is included
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Circuit Access Patency | 12 Months
  Circuit Access Patency is lost when AVF/AVG is intervened on
Primary Assisted Patency | 12 months
  Primary Assisted Patency is lost when circuit undergoes thrombectromy/thrombolysis
Secondary Patency | 12 months
  Secondary Patency is lost when entire dialysis access circuit is abandoned.

CONTACTS AND LOCATIONS:
Overall Officials: Tang Tjun Yip, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No